CLINICAL TRIAL: NCT06776497
Title: The Effect of Vıdeo Streaming with Vırtual Realıty Glasses Durıng Arterıovenous Fıstula Needle Insertıonon on Paın and Anxıety of Indıvıduals Undergoıng Haemodıalysıs Treatment
Brief Title: The Effect of Video Streaming with Virtual Reality Glasses on Pain and Anxiety
Acronym: Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk Ozturk (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Sponsor-Investigator, Selcuk Ozturk, Student, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ERU-SBF-SS-38
Record Dates: First submitted 2024-12-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-03

CONDITIONS: Anxiety; Pain
Keywords: Anxiety; Hemodialysis; Virtual reality glasses; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized, controlled experimental clinical trial to determine the effectiveness of a video played with virtual reality glasseson pain at the vascular access site and anxiety during an AVF catheter procedure in individuals who were undergoing haemodialysis treatment.
Masking Description: No masking done
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- intervention (Experimental): The AVF catheter was inserted into the patients in the virtual reality group just before the clinic's standard haemodialysis procedure (5 minutes earlier), and the video continued to be played until the end of ten minutes after they were connected to the haemodialysis machine. Five minutes after the individual began watching the video, a routine AVF procedure was performed while the individual was still watching the video. During the haemodialysis, the patients in the VRGgroup were allowed to watch videos that they wanted to watch, such as walking in parks, nature and seaside hikes, underwater, museum tours, and feature films with VRGfor 10 minutes. After the time was up, the virtual reality application was terminated, and the VAS and the State-Trait Anxiety Inventory were filled out.
  Interventions: Device: VIRTUAL REALITY GLASSES (VRG)
- control (No Intervention): The control group was subjected to AVF catheter insertion for the standard haemodialysis procedure of the clinic. According to this standard practice, the patients were not subjected to any procedure before AVF access. After they were connected to the haemodialysis machine, the VAS and the StateTrait Anxiety Inventory were completed.

INTERVENTIONS:
Device: VIRTUAL REALITY GLASSES (VRG) — Individuals who met the inclusion criteria and signed the informed consent form were assigned to the study groups based on a list which was numbered and generated in the computer environment before the arteriovenous fistula (AVF) procedure. According to the results given by the computer programme, the individuals were assigned to the control group and the virtual realitiy group (VRG)group. While the control group included patients who underwent AVF procedure with the standard method, the virtual reality headset group included patients who underwent AVF procedure during the VRG application.
  Arms: intervention

SUMMARY:
This study was conducted to examine the effect of a video played with VRG during arteriovenous fistula needle insertionon pain and anxiety of patients undergoing haemodialysis treatment. The sample of the study consisted of a total of 80 patients including 40 in the interventiongroup and 40 in control group who were treated in the haemodialysis ward. The data were collected using aPersonal Information Form prepared by the researcher upon review of the relevant literature to identify the patient's descriptive and medical characteristics, the Visual Analogue Scale (VAS) to assess the severity of pain, and the State-Trait Anxiety Inventory to determine the level of anxiety and VRH.

DETAILED DESCRIPTION:
The data were collected using a Patient Information Form prepared by the researcher upon review of the relevant literature to identify the patient's descriptive and medical characteristics, the Visual Analogue Scale (VAS) to assess the severity of pain, and the State-Trait Anxiety Inventory to determine the level of anxiety and VRH. Additionally, the "Informed Voluntary Consent Form" was used to inform the participants about the study and obtain their consent Individuals who met the inclusion criteria and signed the informed consent form were assigned to the study groups based on a list which was numbered and generated in the computer environment before the AVF procedure. According to the results given by the computer programme, the individuals were assigned to the control group and the VRGgroup.While the control group included patients who

1 2 3 4 5 6 7 8 9 10 11 12 13 14 15 16 17 18 19 20 21 22 23 24 25 26 27 28 29 30 31 32 33 34 35 36 37 38 39 40 41 42 43 44 45 46 47 48 49 50 51 52 53 54 55 56 57 58 59 60 61 62 63 64 65 underwent AVF procedure with the standard method, the virtual reality glasses group included patients who underwent AVF procedure during the VRGapplication. Nurses working in the haemodialysisunit at the time of the study performed AVF procedures in accordance with the haemodialysis procedure protocol. The researcher filled in the descriptive data of the individuals using patient and file records.The individuals were informed about the VAS and the State-Trait Anxiety Inventory.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 18 years and older,
* Those who were not pregnant and had no plans to become pregnant,
* Those who had been undergoing HD treatment in HD wards for at least three months and three sessions per week,
* Those who continued dialysis treatment at the same institution,
* Those for whom there were no changes in the treatment programme during the research period,
* Those who had no pain in any part of the body that would affect the study outcome and scored zero on the Visual Analogue Scale for pain at the time of admission,
* Those who had not taken analgesics in the last 24 hours,
* Those who could understand and communicate in Turkish,
* Those who volunteered to participate in the study and signed the written informed consent form were included in the study.

Exclusion Criteria:

* Those who declined to participate in the study,
* Those with a diagnosed neurological disease such as epilepsy, Alzheimer's disease, Parkinson's disease,and Multiple Sclerosis.
* Those with visual and hearing impairments,
* Those who took anxiolytic and/or sedative medications,
* Those who were clinically unstable,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
The Visual Analogue Scale (VAS) | one week
  The Visual Analogue Scale (VAS) is a tool used to assess the severity of pain. The visual analog scale is a pain rating scale first used by Hayes and Patterson in 1921. It is used to quantify pain that cannot be measured numerically. Two extreme definitions of the pain parameter are written on the two ends of a 100-mm strip, and the patient is asked to indicate where his or her condition fits on this strip by drawing a line, dotting, or marking. It was also found that this scale was easy to understand and applicable for patients over five years of age and was a successful method for assessing the effectiveness of the pain relief method applied. It is a 100-mm (10-cm) ruler that can be used either horizontally or vertically, with no pain at one end and the worst pain at the other end."0 mm" indicates no pain, and "100 mm" indicates the worst pain. The individual indicates the severity of pain felt on this ruler. Based on these data, the horizontally prepared VAS was used to identify th
State-Trait Anxiety Inventory | one week
  State-Trait Anxiety Inventory was developed by Spielberger et al., to assess state and trait anxiety levels and adapted into Turkish by Öner and Lecompte.The scale is based on the two-factor anxiety concept. The Kuder-Richardson reliability of the inventory was found to range from 83 to 87 for the trait anxiety subscale and 94 to 96 for the state anxiety subscale.
  The test-retest reliability rates of the inventory ranged from 71 to 86 for the trait anxiety subscale and from 26 to 68 for the State Anxiety subscale and were considered adequate.In this study, Cronbach's alpha reliability coefficient of the State-Trait Anxiety Inventory was found to be 0.73 for the State Anxiety Inventory and 0.75 for the Trait Anxiety Inventory. The State-Trait Anxiety Inventory consists of a total of 40 items. The first 20 items assess the state-related anxiety level, while the items from 21 to 40 assess the trait anxiety level of the individual.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes Üniversty, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
there is no plan

REFERENCES:
- [Derived] Guler S, Ozturk S, Sahan S, Topaloglu US. The Effect of Video Streaming With Virtual Reality Glasses During Arteriovenous Fistula Needle Insertion on Pain and Anxiety of Individuals Undergoing Hemodialysis Treatment. Hemodial Int. 2025 Jul 24. doi: 10.1111/hdi.70010. Online ahead of print. PMID 40702947